CLINICAL TRIAL: NCT03867916
Title: The Patient Cancer OUtreach, Navigation, Technology, and Support (Patient COUNTS) Project: Addressing Care for Asian Americans With Cancer
Brief Title: Patient Portal and Navigation Program in Providing Information for Asian American Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 184511; NCI-2018-02196 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-03-06; First posted 2019-03-08 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Caregiver; Malignant Neoplasm; Physician; Stage I Colorectal Cancer AJCC v8; Stage I Liver Cancer; Stage I Lung Cancer AJCC v8; Stage IA1 Lung Cancer AJCC v8; Stage IA2 Lung Cancer AJCC v8; Stage IA3 Lung Cancer AJCC v8; Stage IB Lung Cancer AJCC v8; Stage II Colorectal Cancer AJCC v8; Stage II Liver Cancer; Stage II Lung Cancer AJCC v8; Stage IIA Colorectal Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Colorectal Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8; Stage IIC Colorectal Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage III Liver Cancer; Stage III Lung Cancer AJCC v8; Stage IIIA Colorectal Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Colorectal Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms; Liver Neoplasms; Lung Neoplasms | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Health services research (Patient COUNTS) (Experimental): Patients attend focus groups to help develop patient portal and navigation program. Patients use in-person navigation program. Patients also complete data collection and surveys over 15 minutes via web portal at baseline, 3 months, and 6 months and user experience survey at end of program participation.
  Interventions: Behavioral: Patient Navigation Program; Other: Quality-of-Life Assessment; Other: Survey Administration

INTERVENTIONS:
Behavioral: Patient Navigation Program — Use patient navigation program
  Other Names: Patient Navigator Program
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase I/II trial studies how well patient portal and navigation program work in providing information for Asian American cancer patients. Patient portal and navigation program may help to improve the care provided to Asian American cancer patients.This study is offered in the following languages in addition to English: Chinese (Cantonese or Mandarin) and Vietnamese.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identify Asian American adults newly diagnosed with colorectal, liver, or lung cancer using a population-based cancer registry.

II. Conduct outreach to these patients to let them know about the availability of information on these cancers, the Patient Cancer OUtreach, Navigation, Technology and Support (COUNTS) web portal, and the Patient COUNTS patient navigation program.

III. Provide patient navigation either virtually or in-person.

OUTLINE:

Patients attend focus groups to help develop patient portal and navigation program. Patients use in-person navigation program. In phase II, patients use an online portal to access navigation program and may choose to have online/virtual navigation support or in-person navigation support. Patients also complete data collection and surveys over 15 minutes via web portal at baseline, 3 months, and 6 months and user experience survey at end of program participation.

ELIGIBILITY:
Inclusion Criteria:

* FOR INTERVIEWS AND FOCUS GROUPS:

  * Cancer patients: Self-identifies as Asian American, lives in San Francisco, speaks English, Mandarin, Cantonese, or Vietnamese, has a history of cancer of any kind
  * Caregivers: any person age 21 and older who has provided care to an Asian American cancer patient
  * Health professionals: physicians and other health professionals age 21 and older who provide care to Asian American patients with cancer
* FOR PILOT IMPLEMENTATION:

  * Self-identifies as Asian American
  * Ages 21 or older
  * Lives in the 9 counties of the greater bay area cancer registry (GBACR)
  * Speaks English, Mandarin, Cantonese, or Vietnamese
  * Has any stage colorectal, lung, or liver cancer
  * Has not started treatment or has not completed treatment
  * Is willing to stay in the study for six months.
* FOR FULL IMPLEMENTATION:

  * Self-identifies as Asian American
  * Ages 21 or older
  * Lives in the 9 counties of the GBACR
  * Speaks English, Mandarin, Cantonese, or Vietnamese
  * Has any stage colorectal, lung, or liver cancer,
  * Has not started or has not completed treatment
  * Is willing to stay in the study for six-seven months

Exclusion Criteria:

*Any medical or psychological conditions precluding informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of Participation | Any time between consent and month 6
  At least one contact with patient navigator

SECONDARY OUTCOMES:
Adherence to Guideline Treatment | Month 6
  Positive response(s) to survey item(s) on completion of MD-recommended treatment
Patient Acceptability | Month 7
  Response of "satisfied" or "very satisfied" to survey item on satisfaction with Patient COUNTS navigation program

CONTACTS AND LOCATIONS:
Overall Officials: Tung T Nguyen, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang K, Chu JN, Oh DL, Shariff-Marco S, Allen L, Kuo MC, Wong C, Bui H, Chen J, Li FM, Ma C, Truong A, Gomez SL, Nguyen TT, Tsoh JY. Correlates of supportive care needs among Asian Americans with colorectal, liver, or lung cancer from a web-based patient navigation portal intervention: The Patient COUNTS study. Cancer Rep (Hoboken). 2024 Feb;7(2):e1971. doi: 10.1002/cnr2.1971. PMID 38351528
- [Derived] Wang K, Ma C, Li FM, Truong A, Shariff-Marco S, Chu JN, Oh DL, Allen L, Kuo MC, Wong C, Bui H, Chen J, Gomez SL, Nguyen TT, Tsoh JY. Patient-reported supportive care needs among Asian American cancer patients. Support Care Cancer. 2022 Nov;30(11):9163-9170. doi: 10.1007/s00520-022-07338-2. Epub 2022 Aug 30. PMID 36040670